CLINICAL TRIAL: NCT01885195
Title: Modular Phase II Study to Link Targeted Therapy to Patients With Pathway Activated Tumors: Module 3 - MEK162 for Patients With RAS/RAF/MEK Activated Tumors
Brief Title: MEK162 for Patients With RAS/RAF/MEK Activated Tumors
Acronym: SIGNATURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CMEK162AUS11; C4211007 (Other: Alias Study Number)
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Solid Tumor and Hematologic Malignancies
Keywords: RAS, RAF, MEK, NF1, MEK162, signature, papillary thyroid, small intestine, bladder, esophagus, lung cancer, NSCLC, acute myelogenous leukemia, AML
MeSH Terms: conditions — Hematologic Neoplasms; Noonan Syndrome 5; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Leukemia, Myeloid, Acute | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEK162 (Experimental): MEK162 will be dosed on a flat scale of 45 mg twice daily on a continuous dosing schedule.
  Interventions: Drug: MEK162

INTERVENTIONS:
Drug: MEK162 — MEK162 will be dosed on a flat scale of 45 mg twice daily on a continuous dosing schedule.

SUMMARY:
The purpose of this signal seeking study is to determine whether treatment with MEK162 demonstrates sufficient efficacy in select pathway-activated solid tumors and/or hematologic malignancies to warrant further study

DETAILED DESCRIPTION:
This is a phase II, open label study to determine the efficacy and safety of treatment with MEK162 in patients with a diagnosis of select solid tumors or hematological malignancies that have been pre-identified (prior to study consent) to have activations of the RAS/RAF/MEK pathway and whose disease has progressed on or after standard treatment.

Genomic profiling is becoming more accessible to patients and their physicians. This is a signal-seeking study to match patients with mutations in RAF, RAS, NF1 or MEK to the ATP-noncompetitive MEK 1/2 inhibitor, MEK162. Pre-identification of these mutations or activations in the pathway will be performed locally at a CLIA certified laboratory prior to screening for participation on the trial.

Once the patient has been identified, treating physicians who are qualified investigators may contact Novartis to consider enrollment in this study. For the purpose of this study, genomic profiling is not considered part of screening. Informed consent must be signed before any screening activities take place. Once eligibility (screening criteria met) has been confirmed by Novartis, the patient will initiate therapy with single agent MEK162. The patient may not receive any additional anti-cancer therapy during treatment with MEK162.

Patients will continue to receive study treatment until disease progression (assessed by RECIST 1.1 or appropriate hematologic response criteria), unacceptable toxicity, death or discontinuation from study treatment for any other reason (e.g., withdrawal of consent, start of a new anti-neoplastic therapy or at the discretion of the investigator), otherwise known as End of Treatment. All patients who discontinue from study treatment due to disease progression must have their progression clearly documented.

Disease assessment (per RECIST 1.1 or appropriate hematological response criteria) will be performed every 8 weeks (±4 days) after first dose of study drug (Day 1 of every odd cycle), until disease progression or end of treatment, whichever occurs first. The frequency of disease assessment may be reduced to every 12 weeks for patients who have at least 4 post-baseline disease assessments and are clinically stable (except AML and MM patients). Scans will be assessed locally by the investigator. After discontinuation of treatment, patients, regardless of reason for treatment discontinuation, will be followed for safety for 30 days after the last dose.

All patients will be followed for survival status every 3 months for 2 years after the last patient has enrolled in the study regardless of treatment discontinuation reason (except if consent is withdrawn or patient is lost to follow-up.)

ELIGIBILITY:
Inclusion Criteria:

* Patient has a confirmed diagnosis of a select solid tumor (except for primary diagnosis of pancreatic cancer, biliary cancer, colorectal cancer, low grade serous ovarian cancer, melanoma) or hematologic malignancy (except for primary diagnosis of chronic myelomonocytic leukemia).
* Patients must be pre-identified as having a tumor with a mutation in RAF, RAS, NF1 or MEK at a CLIA certified laboratory
* Patient must have received at least one prior treatment for recurrent, metastatic and /or locally advanced disease and for whom no standard therapy options are anticipated to result in a durable remission.
* Patient must have progressive and measurable disease as per RECIST 1.1. or other appropriate hematological guidelines.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1

Exclusion Criteria:

* Patient has received prior treatment with MEK162.
* Patients with primary CNS tumor or CNS tumor involvement
* History of retinal degenerative disease
* History or current evidence of central serous retinopathy (CSR) or retinal vein occlusion (RVO)
* Any ophthalmopathy visible at screening that would be considered a risk factor for CSR or RVO by the ophthalmologist
* Patients who have neuromuscular disorders that are associated with elevated CK

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (68):
- United States (68):
  - University of South Alabama / Mitchell Cancer Institute Univ South Alabama, Mobile, Alabama
  - Alaska Oncology and Hematology AOH (2), Anchorage, Alaska
  - Arizona Oncology Associates AZ Oncology Assoc., Phoenix, Arizona
  - Arizona Oncology Associates HOPE Division, Phoenix, Arizona
  - Arizona Oncology Associates PC- NAHOA, Sedona, Arizona
  - Highlands Oncology Group Highlands Oncology Group (22), Fayetteville, Arkansas
  - PCR Oncology, Pismo Beach, California
  - University of California Davis Cancer Center UC Davis Cancer (3), Sacramento, California
  - Rocky Mountain Cancer Centers USOR, Boulder, Colorado
  - Yale University School of Medicine Yale Cancer Center, New Haven, Connecticut
  - Whittingham Cancer Center Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology & Oncology Associates Dept. of ECHO, Norwich, Connecticut
  - Hematology Oncology PC Stamford Hospital, Stamford, Connecticut
  - Florida Cancer Specialists Florida Cancer Specialists (31, Fort Myers, Florida
  - Memorial Cancer Institute Memorial Healthcare System, Hollywood, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Mt. Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Ocala Oncology Center Dept. of Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida PA Cancer Centers of FL-Orlando-4, Ocoee, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Lurie Children's Hospital of Chicago Developmental Therapeutics, Chicago, Illinois
  - Oncology Specialists, SC Onc Specialists, Park Ridge, Illinois
  - Illinois Cancer Care IL. Cancer Care, Peoria, Illinois
  - Indiana University Indiana Univ. - Purdue Univ., Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics Regulatory Contact 2, Iowa City, Iowa
  - Maryland Oncology Hematology, P.A. Oncology Hematology, Rockville, Maryland
  - Cancer and Hematology Centers of West Michigan Dept. of Oncology, Grand Rapids, Michigan
  - Metro MN CCOP - Coon Rapids, Coon Rapids, Minnesota
  - Research Medical Center Research Med Center (2), Kansas City, Missouri
  - Washington University School of Medicine Washington University (16), St Louis, Missouri
  - Glacier View Research Institute - Cancer Oncology Dept, Kalispell, Montana
  - Comprehensive Cancer Centers of Nevada CCC of Nevada (21), Las Vegas, Nevada
  - Cancer Institute of New Jersey CINJ, New Brunswick, New Jersey
  - New Mexico Cancer Care Alliance Oncology Dept, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C. NYOH Latham, Troy, New York
  - University of North Carolina Chapel Hill Physician Office Building, Chapel Hill, North Carolina
  - Duke University Medical Center Seeley G. Mudd Bldg., Durham, North Carolina
  - Sanford Research/USD-Fargo Sanford Hematology Oncology, Fargo, North Dakota
  - Cleveland Clinic Foundation Cleveland Clinic (19), Cleveland, Ohio
  - Ohio State University Medical Center Comprehensive Cancer Center, Columbus, Ohio
  - St. Charles Cancer Center, Bend, Oregon
  - Willamette Valley Clinical Studies Cancer Institute & Res. Ctr., Eugene, Oregon
  - Northwest Cancer Specialists Vancouver Cancer Center, Portland, Oregon
  - Oregon Health & Science University Oregon Health & Science U (56), Portland, Oregon
  - St. Luke's Hospital and Health Network St Luke's (2), Bethlehem, Pennsylvania
  - West Penn Allegheny Oncology Network, Natrona Heights, Pennsylvania
  - Abington Hematology Oncology Associates, Inc Abington Hem Onc Assoc (5), Willow Grove, Pennsylvania
  - Chattanooga Oncology and Hematology Assoicates, PC Chattanooga Oncology, Chattanooga, Tennessee
  - The West Clinic Dept. of the West Clinic, Memphis, Tennessee
  - Sarah Cannon Research Institute Sarah Cannon Research Inst (51, Nashville, Tennessee
  - Texas Oncology Presbyterian Hospital (3), Dallas, Texas
  - Texas Oncology Texas Oncology - Denton, Dallas, Texas
  - Texas Oncology Austin Midtown, Dallas, Texas
  - Texas Oncology Texas Oncology - Midland, Dallas, Texas
  - Sammons Cancer Center - Texas Oncology Sammons Cancer Center (10), Dallas, Texas
  - Oncology Consultants Oncology Group, Houston, Texas
  - MD Anderson Cancer Center/University of Texas MD Anderson Cancer Center (3), Houston, Texas
  - Cancer Care Centers of South Texas / HOAST CCC of So. TX-San Antonio (3), San Antonio, Texas
  - Tyler Cancer Center Dept.ofTylerCancerCtr. (2), Tyler, Texas
  - Deke Slayton Cancer Center Deke Slayton Cancer Center (2), Webster, Texas
  - Intermountain Medical Center Intermountain Healthcare, Murray, Utah
  - Virginia Cancer Specialists, PC Virginia Cancer Specialists, Fairfax, Virginia
  - Medical Oncology & Hematology Associates of Northern VA Med Onc Hem Northern VA, Reston, Virginia
  - Kadlec Clinic Hematology and Oncology Kadlec Clinic Hematology & Onc, Kennewick, Washington
  - Providence Regional Cancer System, Lacey, Washington
  - MultiCare Health System Institute for Research & Innovation MultiCare, Tacoma, Washington
  - Northwest Medical Specialties NW Medical Specialties, Tacoma, Washington
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Burkart J, Owen D, Shah MH, Abdel-Misih SRZ, Roychowdhury S, Wesolowski R, Haraldsdottir S, Reeser JW, Samorodnitsky E, Smith A, Konda B. Targeting BRAF Mutations in High-Grade Neuroendocrine Carcinoma of the Colon. J Natl Compr Canc Netw. 2018 Sep;16(9):1035-1040. doi: 10.6004/jnccn.2018.7043. PMID 30181415

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants diagnosed with select solid tumors or hematological malignancies pre-identified (prior to study consent) and had an activation of the v-raf murine sarcoma viral oncogene (RAF)/ RAS oncogene [rat sarcoma viral oncogene homologue] (RAS)/mitogen-activated erk kinase (MEK) pathway and whose disease had progressed on or after standard treatment.
Groups:
- Binimetinib (MEK162): Participants received an oral dose of 45 milligram (mg) of binimetinib tablets (3 tablets of 15 mg) twice daily in each cycle starting from Cycle 1 Day 1 (1 cycle =28 days) until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment due to any other reason. Maximum treatment exposure was approximately of 19.4 months.
Period: Overall Study
Arm/Group | Binimetinib (MEK162)
Started | 110
Completed | 0
Not Completed | 110
Not completed — Adverse Event | 29
Not completed — Death | 1
Not completed — Disease Progression | 67
Not completed — Protocol Deviation | 2
Not completed — Physician Decision | 3
Not completed — Patient/guardian decision | 8

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Binimetinib (MEK162): Participants received an oral dose of 45 mg of binimetinib tablets (3 tablets of 15 mg) twice daily in each cycle starting from Cycle 1 Day 1 (1 cycle =28 days) until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment due to any other reason. Maximum treatment exposure was approximately of 19.4 months.
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) for Solid Tumors at Week 16 as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: CBR: participants with complete response (CR), partial response (PR) or stable disease (SD) for at least 16 weeks. As per RECIST 1.1, CR: disappearance of all target and non-target lesions, normalization of tumor marker level, pathological lymph nodes assigned as target or non-target lesions must have a reduction in short axis to less than (<) 10 millimeter (mm); PR: at least a 30 percent (%) decrease in sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters; PD: at least a 20% increase in sum of diameter of all measured target lesions, taking as reference smallest sum of diameter of all target lesions recorded at or after baseline, sum was also an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. Appearance of >=1 new target or non-target lesions.
Time Frame: Week 16
Population: Full analysis set included all the participants who had received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 104
Percentage of participants | 23.1 [15.4 to 32.4]

2. Primary Outcome: CBR for Hematologic Tumors at Week 16: Multiple Myeloma
Description: CBR: participants with stringent complete response(sCR), CR, very good partial response(VGPR), PR/SD for at least 16 weeks. For hematologic tumors (multiple myeloma), sCR: negative immunofixation on serum, urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow plus normal free light chain(FLC) ratio and absence of clonal cells in bone marrow by immunohistochemistry/immunofluorescence; CR: negative immunofixation on the serum, urine, disappearance of any soft tissue, plasmacytomas and <5% plasma cells in bone marrow; VGPR: serum,urine M-component detectable by immunofixation but not on electrophoresis or>=90% reduction in serum M-component plus urine M-component <100 mg/24 hr; PR: >50% reduction of serum M-protein and reduction in 24hr urinary M-protein by >90%/to <200 mg/24 hr; SD: not meeting criteria for CR, VGPR, PRor PD; PD: increase of >25% from lowest response value in serum M-component, urine M-component and bone marrow plasma cell percentage.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 3
Percentage of participants | 0.0 [0.0 to 70.8]

3. Primary Outcome: CBR for Hematologic Tumors at Week 16: Acute Myeloid Leukemia
Description: CBR: participants with complete remission (CR), CR with incomplete blood count recovery (CRi), partial remission (PR) and no resposne for at least 16 weeks. For hematologic tumors (acute myeloid leukemia); CR: as bone marrow- < 5% blasts, no blasts with auer rods, peripheral blood- neutrophils ≥1.0*10^9/L and/or platelets ≥100*10^9/L, ≤1% blasts, no evidence of extramedullary disease (such as CNS or soft tissue involvement), transfusion independent; CRi: all the CR criteria were involved but platelet and neutrophil transfusions were also allowed; PR: bone marrow- 50% or greater decrease (absolute range 5-25% blasts), < 5% of blasts contain auer rods, peripheral blood- neutrophils <1.0*10^9/L and/or platelets <100*10^9/L, no evidence of extramedullary disease; no response: in case a patient did not achieve CR, CRi, PR or relapse for an individual response assessment.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 3
Percentage of participants | 33.3 [0.8 to 90.6]

4. Secondary Outcome: Overall Response Rate (ORR) as Per RECIST Version 1.1
Description: ORR: percentage of participants with a best overall response (BOR) of CR or PR as assessed per RECIST version 1.1. BOR: the best response recorded from the start of the treatment until disease progression (PD). CR: disappearance of all target and non-target lesions, normalization of tumor marker level, pathological lymph nodes assigned as target or non-target lesions must have a reduction in short axis to less than <10 mm; PR: at least a 30 % decrease in sum of diameter of all target lesions, taking as reference the baseline sum of diameters; PD: at least a 20% increase in sum of diameter of all measured target lesions, taking as reference smallest sum of diameter of all target lesions recorded at or after baseline, sum was also an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. Appearance of >=1 new target or non-target lesions.
Time Frame: From the start of the treatment until disease progression (maximum up to 19.4 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 104
Percentage of participants | 2.9 [0.6 to 8.2]

5. Secondary Outcome: ORR for Hematologic Tumors: Multiple Myeloma
Description: ORR: percentage of participants with sCR, CR, VGPR or PR. For hematologic tumors (multiple myeloma), sCR: negative immunofixation on the serum, urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; CR: CR: negative immunofixation on the serum, urine, disappearance of any soft tissue, plasmacytomas and <5% plasma cells in bone marrow; VGPR: serum and urine M-component detectable by immunofixation but not on electrophoresis or greater than equal to >=90% reduction in serum M-component plus urine M-component <100 mg per 24hour (hr); PR: >50% reduction of serum M-protein and reduction in 24 hr urinary M-protein by >90% or to <200 mg/24 hr.
Time Frame: From the start of the treatment until disease progression (maximum up to 19.4 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 3
Percentage of participants | 33.3 [0.8 to 90.6]

6. Secondary Outcome: ORR for Hematologic Tumors: Acute Myeloid Leukemia
Description: ORR: participants with complete remission (CR), CR with incomplete blood count recovery (CRi), partial remission (PR) and no resposne for at least 16 weeks. For hematologic tumors (acute myeloid leukemia); CR: as bone marrow- < 5% blasts, no blasts with auer rods, peripheral blood- neutrophils ≥1.0*10^9/L and/or platelets ≥100*10^9/L, ≤1% blasts, no evidence of extramedullary disease (such as CNS or soft tissue involvement), transfusion independent; CRi: all the CR criteria were involved but platelet and neutrophil transfusions were also allowed; PR: bone marrow- 50% or greater decrease (absolute range 5-25% blasts), < 5% of blasts contain auer rods, peripheral blood- neutrophils <1.0*10^9/L and/or platelets <100*10^9/L, no evidence of extramedullary disease.
Time Frame: From the start of the treatment until disease progression (maximum up to 19.4 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 3
Percentage of participants | 33.3 [0.8 to 90.6]

7. Secondary Outcome: Progression-free Survival (PFS) as Per RECIST Version 1.1
Description: PFS was defined as the time from the date of first dose to the date of first documented PD or relapse or death due to any cause. PD: at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. Appearance of >=1 new target or non-target lesions was also considered progression. PFS data was censored at date of last adequate tumor assessment.
Time Frame: From the date of first dose to the date of the first documented PD, censored date or death (maximum up to 19.4 months)
Population: Full analysis set included all the participants who had received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 110
Months | 2.6 [1.9 to 3.5]

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to the date of death due to any cause. If a participant was not known to have died, survival time was censored at the date of last contact.
Time Frame: From the date of first dose to the date of death due to any cause (maximum up to 19.4 months)
Population: Full analysis set included all the participants who had received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 110
Months | 8.5 [6.6 to 11.8]

9. Secondary Outcome: Duration of Response (DOR) as Per RECIST Version 1.1
Description: DOR was defined as the time from the first documented response (CR or PR) to the date of first documented disease progression, relapse or death due to any cause. As per RECIST 1.1, CR: disappearance of all target and non-target lesions, normalization of tumor marker level, pathological lymph nodes assigned as target or non-target lesions must have a reduction in short axis to <10 mm; PR: at least a 30% decrease in sum of diameter of all target lesions, taking as reference the baseline sum of diameters; PD: at least a 20% increase in sum of diameter of all measured target lesions, taking as reference smallest sum of diameter of all target lesions recorded at or after baseline, sum was also an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. Appearance of >=1 new target or non-target lesions. The DOR was determined only in participants whose best response was PR or greater.
Time Frame: From the first documented response (CR or PR) to the date of the first documented PD or death (maximum up to 19.4 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 3
Months | NA [NA to NA] — Median and 95% CI were not estimable due to low number of participants who had an event.

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Graded According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical/diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local/noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated. Treatment-emergent adverse events were defined as new or worsening events that were collected from first study treatment date to last treatment date +30 days. AEs of all grades were reported.
Time Frame: From Baseline up to 30 days following the last dose of study treatment (maximum up to 21 months)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment and had at least 1 post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 110
Participants
  Grade 1 | 2
  Grade 2 | 27
  Grade 3 | 64
  Grade 4 | 17

11. Secondary Outcome: Number of Participants With Vital Sign Abnormality of Greater Than or Equal to (>=) Grade 3 as Per CTCAE v4.03
Description: Vital signs included hypertension, hypotension and weight decreased were reported. As per NCI-CTCAE version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical/diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local/noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated. Participants with grade 3 or higher vital sign abnormality are reported.
Time Frame: From Baseline up to 30 days following the last dose of study treatment (maximum up to 21 months)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 110
Participants
  Hypertension | 15
  Hypotension | 6
  Weight Decreased | 11

12. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities criteria included: 1) QTc interval adjusted according to Bazett formula (QTcF) in millisecond (msec): greater than equal to (>=) 450 to less than (<) 480, >=480 to <500, >=500, increase from baseline >=30, increase from baseline >=60; 2) QTc interval adjusted according to Fridericia formula (QTcB) (msec): >=450 to <480, >=480 to <500, >=500, increase from baseline >=30, increase from baseline >=60. 3) QT (msec): >=450 to <480, >=480 to <500, >=500, increase from baseline >=30, increase from baseline >=60.
Time Frame: From Baseline up to 30 days following the last dose of study treatment (maximum up to 21 months)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 110
Participants
  QTcF: >=450 to <480 msec | 15
  QTcF: >=480 to <500 msec | 4
  QTcF: >=500 msec | 1
  QTcF: Increase from baseline >=30 msec | 20
  QTcF: Increase from baseline >=60 msec | 3
  QTcB: >=450 to <480 msec | 13
  QTcB: >=480 to <500 msec | 5
  QTcB: >=500 msec | 8
  QTcB: Increase from baseline >=30 msec | 53
  QTcB: Increase from baseline >=60 msec | 29
  QT: >=450 to <480 msec | 13
  QT: >=480 to <500 msec | 2
  QT: >=500 msec | 2
  QT: Increase from baseline >=30 msec | 39
  QT: Increase from baseline >=60 msec | 7

13. Secondary Outcome: Number of Participants With Shift From Baseline in Clinical Laboratory - Hematology Parameters
Description: Laboratory parameters included hematological and biochemistry parameters. Hematological parameters included neutrophils, platelets, prothrombin time, activated partial thromboplastin time, INR, fibrinogen. Number of participants with hematological abnormalities by grades (as per Common Terminology Criteria for Adverse Events (CTCAE version 4.03) were reported. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Participants with a grade shift of 3 or more from baseline are reported in this outcome measure.
Time Frame: From Baseline up to 30 days following the last dose of study treatment (maximum up to 21 months)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment and had at least 1 post-baseline safety assessment. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 110
Participants
  Neutrophils: number analyzed (Participants) | 85
  Neutrophils | 6
  Platelets: number analyzed (Participants) | 77
  Platelets | 3
  Prothrombin Time: number analyzed (Participants) | 73
  Prothrombin Time | 2
  Activated Partial Thromboplastin Time: number analyzed (Participants) | 69
  Activated Partial Thromboplastin Time | 2
  INR: number analyzed (Participants) | 80
  INR | 2
  Fibrinogen: number analyzed (Participants) | 81
  Fibrinogen | 0

14. Secondary Outcome: Number of Participants With Shift From Baseline in Clinical Laboratory - Biochemistry Parameters
Description: Laboratory parameters included hematological and biochemistry parameters. Biochemistry parameters included: creatinine, phosphorus, albumin, gamma-glutamyl transferase, aspartate transaminase, alanine aminotransferase, alkaline phosphatase, total bilirubin, uric acid, amylase, lipase, creatine kinase, total cholesterol and triglycerides. Number of participants with biochemistry test abnormalities by grades (CTCAE version 4.03) were reported. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Participants with a grade shift of 3 or more from baseline are reported in this outcome measure.
Time Frame: From Baseline up to 30 days following the last dose of study treatment (maximum up to 21 months)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 110
Participants
  Creatinine: number analyzed (Participants) | 81
  Creatinine | 0
  Phosphorus: number analyzed (Participants) | 98
  Phosphorus | 1
  Albumin: number analyzed (Participants) | 33
  Albumin | 5
  Gamma-Glutamyl Transferase: number analyzed (Participants) | 68
  Gamma-Glutamyl Transferase | 1
  Aspartate Transaminase: number analyzed (Participants) | 39
  Aspartate Transaminase | 2
  Alanine Aminotransferase: number analyzed (Participants) | 76
  Alanine Aminotransferase | 2
  Alkaline Phosphatase: number analyzed (Participants) | 58
  Alkaline Phosphatase | 0
  Total Bilirubin: number analyzed (Participants) | 104
  Total Bilirubin | 0
  Uric Acid: number analyzed (Participants) | 91
  Uric Acid | 0
  Amylase: number analyzed (Participants) | 81
  Amylase | 2
  Lipase: number analyzed (Participants) | 85
  Lipase | 5
  Creatine Kinase: number analyzed (Participants) | 28
  Creatine Kinase | 18
  Total Cholesterol: number analyzed (Participants) | 73
  Total Cholesterol | 0
  Triglycerides: number analyzed (Participants) | 59
  Triglycerides | 1

15. Secondary Outcome: Number of Participants With Shift From Baseline in Cardiac Imaging
Description: Number of Participants With Shift From Baseline in Cardiac Imaging were reported.
Time Frame: From Baseline up to 30 days following the last dose of study treatment (maximum up to 21 months)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 110
Participants | 10

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days following the last dose of study treatment (maximum up to 21 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis set included all the participants who received at least 1 dose of study treatment and had at least 1 post-baseline safety assessment.
Arm/Group | Binimetinib (MEK162)
Serious Adverse Events (participants affected / at risk) | 50/110
Other Adverse Events (participants affected / at risk) | 110/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Binimetinib (MEK162) (N=110)
Coagulopathy (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Dilatation ventricular (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Retinal artery occlusion (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Retinal tear (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Small intestinal obstruction (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1
Oesophageal perforation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 2
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Bile duct obstruction (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Troponin I increased (Investigations) | 1
Troponin T increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Lymphorrhoea (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Binimetinib (MEK162) (N=110)
Anaemia (Blood and lymphatic system disorders) | 29
Neutropenia (Blood and lymphatic system disorders) | 7
Vision blurred (Eye disorders) | 18
Chorioretinopathy (Eye disorders) | 8
Periorbital oedema (Eye disorders) | 7
Visual impairment (Eye disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 52
Nausea (Gastrointestinal disorders) | 48
Vomiting (Gastrointestinal disorders) | 42
Constipation (Gastrointestinal disorders) | 25
Dry mouth (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 55
Oedema peripheral (General disorders) | 44
Mucosal inflammation (General disorders) | 13
Pyrexia (General disorders) | 13
Asthenia (General disorders) | 11
Face oedema (General disorders) | 10
Chills (General disorders) | 7
Oedema (General disorders) | 7
Urinary tract infection (Infections and infestations) | 19
Blood creatine phosphokinase increased (Investigations) | 38
Aspartate aminotransferase increased (Investigations) | 22
Alanine aminotransferase increased (Investigations) | 15
Lipase increased (Investigations) | 13
Amylase increased (Investigations) | 11
Blood lactate dehydrogenase increased (Investigations) | 11
Ejection fraction decreased (Investigations) | 11
Weight decreased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 9
Blood phosphorus increased (Investigations) | 8
Blood creatinine increased (Investigations) | 6
Gamma-glutamyltransferase increased (Investigations) | 6
Intraocular pressure increased (Investigations) | 6
Troponin T increased (Investigations) | 6
White blood cell count decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 24
Hypomagnesaemia (Metabolism and nutrition disorders) | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 14
Dehydration (Metabolism and nutrition disorders) | 11
Hypokalaemia (Metabolism and nutrition disorders) | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 7
Neuropathy peripheral (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 10
Anxiety (Psychiatric disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 48
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 21
Dry skin (Skin and subcutaneous tissue disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Hypertension (Vascular disorders) | 15
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.